CLINICAL TRIAL: NCT03477708
Title: The Impact of Continuous Transcutaneous CO2 Monitoring (TCCO2) in Extremely Low Birth Weight (ELBW) Infants: A Prospective Observational, Multi-Center Study
Brief Title: The Impact of Continuous Transcutaneous CO2 (TCCO2) Monitoring in Extremely Low Birth Weight (ELBW) Infants
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Liron Borenstein MD, Liron Borenstein Levin,MD, Neonatologist, Rambam Health Care Campus
Other Study IDs: TCCO2 monitoring in ELBW
Record Dates: First submitted 2018-03-07; First posted 2018-03-26 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: ELBW - Extremely Low Birth Weight Infant; IVH- Intraventricular Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: TCCO2 monitoring
- Control group: Routine monitoring

SUMMARY:
An observational study comparing outcomes of Extremely Low Birth Weight (ELBW) infants that were monitored with non-invasive Transcutaneous CO2 (TCCO2) monitor to infants that were not monitored by TCCO2 monitor.

ELIGIBILITY:
Inclusion Criteria:

* ELBW infants Need of respiratory support

Exclusion Criteria:

* Parental refusal IVH before study entry chromosomal abnormalities congenital central nervous system (CNS) abnormalities

Ages: 0 Minutes to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ELBW infants
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
IVH-Intraventricular Hemorrhage | Repeated scans until infant reaches corrected age of 42 weeks
  Intraventricular Hemorrhage
PVL- Periventricular Leukomalacia | Repeated scans until infant reaches corrected age of 42 weeks
  Periventricular Leukomalacia

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No